CLINICAL TRIAL: NCT00251277
Title: Use of Rituximab Treatment in Addition to Standard Care for Newly Presenting Thrombotic Thrombocytopenic Purpura
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, James B. Bussel, Professor of pediatrics, Weill Medical College of Cornell University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0409007463
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: Thrombotic Thrombocytopenic Purpura; TTP; Hematology
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rituximab — Rituximab will be administered immediately after pheresis to minimize the amount of Rituximab that is removed by the subsequent days pheresis. The guidelines will be that 12 hours must elapse between the end of the first infusion of study drug and the next pheresis. Subsequent infusions would be weekly (plus or minus 2 days) with an attempt made to give study drug infusions after a pheresis that might be the last in a series, i.e. when no pheresis would be scheduled for at least the next day.

SUMMARY:
The purpose is to evaluate safety and feasibility of the use of Rituximab as an adjunct to standard therapy (plasmapheresis + steroids) for patients with thrombotic thrombocytopenic purpura (TTP). This includes evaluating the rate and type of treatment failure.

DETAILED DESCRIPTION:
With this study we hope to evaluate safety and feasibility of the use of Rituximab as an adjunct to standard therapy (plasmapheresis + steroids) for patients with thrombotic thrombocytopenic purpura (TTP). This includes evaluating the rate and type of treatment failure.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the trial based on the following criteria:

* Patients must have TTP with platelet count < 100,000/mL and microangiopathic hemolytic anemia which is defined as presence of at 3-10 fragmented red blood cells (schistocytes) per high power filed on the peripheral blood smear.
* Either gender, age 17 or older
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* TTP not related to underlying cancer, treatment of cancer or transplantation
* New onset TTP, or previously diagnosed TTP with an unmaintained remission for >12 months.
* LDH >2X upper limit of normal
* Prothrombin time (PT), partial thromboplastin time (PTT) normal
* Direct antiglobulin test (DAT) negative
* Subject has provided written informed consent
* Patients who have received up to 3 plasmapheresis.

Exclusion Criteria:

Patients will be excluded from the trial based on the following criteria:

* A diagnosis of AIDS. Patients with HIV infection with absolute CD4 counts >200/ul and no active, significant opportunistic infection are eligible
* Patients with a known hepatitis C infection (HCV) and/or with hepatitis B
* Patients receiving pheresis more than once a day
* Recent (within 1 year) bone marrow or hematopoietic stem cell transplant
* Patient is on calcineurin inhibitors, or is unable to come off them
* Acute or chronic disseminated intravascular coagulation (DIC), defined by D-dimers >8mg/ml and fibrinogen < 100 mg (0.1g)/dl
* A diagnosis of metastatic or non-metastatic malignancy other than basal cell carcinoma.
* Malignant hypertension (systolic blood pressure [BP] > 200 mm Hg or a diastolic BP > 130 mm Hg)
* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment). Eligibility resumes 3 days after delivery
* Patients with family history of or a previous diagnosis of congenital TTP
* Patients with hemolytic uremic syndrome (HUS)
* Patients with sepsis

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Failure to maintain the complete response until day 120; Non-protocol treatment for TTP, such as other immunosuppressive agents or splenectomy, reinstitution of plasma exchange within the first 90 days | Four months

CONTACTS AND LOCATIONS:
Overall Officials: James B Bussel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University/New York Presbyterian Hospital, New York, New York, United States